CLINICAL TRIAL: NCT00086372
Title: Acute HIV Infection and Early Disease Research Program (AIEDRP) CORE01 Database
Brief Title: Long-term Follow-up of HIV Infected Patients Identified During Early Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); Acute Infection and Early Disease Research Program (Network)
Responsible Party: Sponsor
Other Study IDs: AIEDRP CORE01; ACTG A5228
Record Dates: First submitted 2004-06-30; First posted 2004-07-01 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections

SUMMARY:
This is a long-term follow-up study of people who are identified during acute or recent HIV infection and are being followed at clinical research sites associated with the Acute HIV Infection and Early Disease Research Program (AIEDRP).

DETAILED DESCRIPTION:
AIEDRP was established to develop and evaluate data from studies of patients with acute or recent HIV infection. Long-term effects of antiretroviral therapies raise questions regarding the value and necessity of therapeutic interventions during acute and early HIV infection. Conventional randomized clinical trials are generally designed with finite endpoints; most patients who reach an endpoint or complete a protocol are no longer followed. As a result, long-term virologic, immunologic, and clinical outcome data are not available. This is particularly true for participants who fail therapy, require changes in treatment, or develop a treatment-limiting toxicity in a time-limited study.

This database study will establish a cohort of HIV infected individuals who are participating in HIV studies at AIEDRP sites and of HIV infected individuals who have chosen to defer therapy but agree to be followed by this study. The study will facilitate longitudinal and prospectively planned meta-analyses or cross-protocol analyses of AIEDRP studies by developing data collection guidelines, defining common research goals, and creating data templates. The primary aim is to determine the long-term virologic, immunologic, and clinical outcomes and complications for patients who were diagnosed during acute or early HIV infection.

Participants in this study will be followed for at least 5 years. Study visits will occur at Weeks 2, 4, and 12, and then every 12 weeks thereafter, through Week 96. After 2 years, study visits will occur every 24 weeks until the end of the study. Participants who start antiretroviral therapy at or after Week 2 will restart the study visit schedule. Study visits will include a medical interview, adherence questionnaire, and blood tests. Duplicate tests performed as part of another study will not be performed if the results of those tests are available.

ELIGIBILITY:
Inclusion Criteria

* Documented acute or recent HIV infection
* Willing to allow study investigators access to and use of participant's medical information from other AIEDRP clinical trials
* Parent or guardian willing to provide informed consent, if applicable
* If enrolled at an AIDS Clinical Trial Group (ACTG) site, must also be participating in one of the following clinical trials: AIN501/ACTG A5216, AIN503/ACTG A5217, or AIN504/ACTG A5218

Exclusion Criteria

* More than 7 days of antiretroviral therapy prior to study entry without adequate documentation of pretreatment viral load and CD4 count. Individuals who have failed postexposure prophylaxis with antiretroviral treatment are not excluded from enrollment.
* Any factor that, in the opinion of the study official, may interfere with study participation

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2003-07; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Study Chair — Aaron Diamond AIDS Research Center, Rockefeller University; Susan Little, MD, Study Chair — University of California, San Diego
Locations (30):
- United States (22):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Cedars-Sinai, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts
  - Community Research Initiative of New England-Sprin, Springfield, Massachusetts
  - Washington University (St. Louis), St Louis, Missouri
  - State University of NY Downstate, Brooklyn, New York
  - Beth Israel Medical Center, New York, New York
  - Aaron Diamond AIDS Research Center, New York, New York
  - Columbia University, New York, New York
  - Community Health Network, Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Presbyterian Medical Center - Univ. of PA, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Australia (4):
  - University of New South Wales, Darlinghurst, New South Wales
  - Prahran Market Clinic, St Kilda, Victoria
  - The Centre Clinic, St Kilda, Victoria
  - Carlton Clinic, Carlton VID
- Centro de Referencia Estadual de AIDS (CREAIDS), Salvador, Estado de Bahia, Brazil
- Canada (2):
  - University of British Columbia, Vancouver, BC, Vancouver, British Columbia
  - Montreal Chest Institute of the McGill University, Montreal, Quebec
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

REFERENCES:
- [Background] Kassutto S, Rosenberg ES. Primary HIV type 1 infection. Clin Infect Dis. 2004 May 15;38(10):1447-53. doi: 10.1086/420745. Epub 2004 Apr 30. PMID 15156484
- [Background] Pilcher CD, Eron JJ Jr, Galvin S, Gay C, Cohen MS. Acute HIV revisited: new opportunities for treatment and prevention. J Clin Invest. 2004 Apr;113(7):937-45. doi: 10.1172/JCI21540. PMID 15057296
- [Result] Falster K, Gelgor L, Shaik A, Zablotska I, Prestage G, Grierson J, Thorpe R, Pitts M, Anderson J, Chuah J, Mulhall B, Petoumenos K, Kelleher A, Law M. Trends in antiretroviral treatment use and treatment response in three Australian states in the first decade of combination antiretroviral treatment. Sex Health. 2008 Jun;5(2):141-54. doi: 10.1071/sh07082. PMID 18588779